CLINICAL TRIAL: NCT02958215
Title: A Study Evaluating Hypotension and Autonomic Nervous System Dysfunction During Spinal Anesthesia for Cesarean Section and Its Relation to the Effect of Prophylaxis Phenylephrine
Brief Title: Phenylephrine and Hypotension During Spinal Anesthesia for Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate profossor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB0000871230
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Anesthesia, Obstetrical; Anesthesia, Spinal
Keywords: Orthostatic; Cesarean section; Pregnant; Phenyephrine; Hypotension
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Placebo Comparator): This group will include patients with orthostatic hypotension and will be managed with routine spinal anesthesia Ephedrine will be used for management of intraoperative hypotension
  Interventions: Other: Placebo
- Group B (Active Comparator): This group will include patients with orthostatic hypotension and will be managed with prophylaxis single dose of phenylephrine, 50 ug IV, will be administered immediately before the spinal block then the patients will be managed with routine spinal anesthesia Ephedrine will be used for management of intraoperative hypotension
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine — it will be given as a prophylaxis for prevention of hypotension after spinal anesthesia in pregnant patients undergoing cesarean section
  Arms: Group B
Other: Placebo — 5 ml normal saline will be given before spinal anesthesia
  Arms: Group A

SUMMARY:
Pregnant women with a positive preoperative Supine stress test were found to be a subgroup at increased risk of symptomatic hypotension after spinal anesthesia

DETAILED DESCRIPTION:
Patients will be placed in dorsal decubitus dislocating the uterus to the left for a few minutes, with blood pressure and heart rate recorded three times, with a three-minute interval between measurements to obtain mean baseline levels and this will be repeated in an upright position to record the same measurement.Orthostatic hypotension (Orthostatic hypotension "OH" is defined specifically as a 20mmHg drop in systolic, and/or a 10mmHg drop in diastolic blood pressure within 3 minutes of standing.

ELIGIBILITY:
Inclusion Criteria:

Physical status ASA I, A full term pregnancy A single fetus Elective cesarean section.

Exclusion Criteria:

Refusal of the patient to participate in the study History of hypertension Pregnancy-induced hypertension Cardiovascular or cerebrovascular disease Fetal abnormalities History of hypersensitivity to the drugs used Contraindications to spinal block.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 980 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | within first 24 hours after spinal anesthesia
  blood pressure will be measured every 3 minutes within the first 30 minutes after spinal block the every 5 minutes till the end of the caesarian section. postoperatively will be checked every 15 minutes in the first hour the every 30 minutes till the recovery from spinal block

SECONDARY OUTCOMES:
Frequency of bradycardia | within first 24 hours after spinal anesthesia
  heart rate will be measured every 5 minutes till the end of the caesarian section. postoperatively will be checked every 15 minutes in the first hour the every 30 minutes till the recovery from spinal block
Ephedrine usage | within first 24 hours after spinal anesthesia
  Total amount of ephedrine given
intraoperative fluid management | within first 24 hours after spinal anesthesia
  Total amount of fluid given
Apgar scores | within first 24 hours after spinal anesthesia
  Apgar scores in the first and fifth minutes of the newborns

CONTACTS AND LOCATIONS:
Overall Officials: Sayed K Abd-Elshafy, MD, Principal Investigator — Associate professor of anesthesia
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided